CLINICAL TRIAL: NCT03697941
Title: Percutaneous Plug-based Arteriotomy Closure Device Use in Minimally Invasive Mitral Valve Surgery
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Dalén, MD, PhD, Karolinska University Hospital
Other Study IDs: MIMVS-MANTA
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical cut-down and arterial puncture under direct vision
  Interventions: Procedure: Surgical cut-down and arterial puncture under direct vision
- Percutaneous arteriotomy closed with closure device
  Interventions: Procedure: Percutaneous arteriotomy closed using a plug-based arteriotomy closure device

INTERVENTIONS:
Procedure: Percutaneous arteriotomy closed using a plug-based arteriotomy closure device — Percutaneous arteriotomy closed using a plug-based arteriotomy closure device (MANTA, Essential Medical Inc., Malvern, Pennsylvania).
  Groups: Percutaneous arteriotomy closed with closure device
Procedure: Surgical cut-down and arterial puncture under direct vision — Surgical cut-down and arterial puncture under direct vision.
  Groups: Surgical cut-down and arterial puncture under direct vision

SUMMARY:
A single-center prospective study. Patients undergoing minimally invasive mitral valve surgery between February 2016 and December 2018 at the Karolinska University Hospital in Stockholm, Sweden are eligible. Femoral cannulation was performed either with surgical cut-down and arterial puncture under direct vision or percutaneously with planned percutaneous arteriotomy closed using a plug-based arteriotomy closure device (MANTA, Essential Medical Inc., Malvern, Pennsylvania). Data regarding preoperative clinical characteristics and operative details were obtained by medical records review and from the Swedish Web system for Enhancement and Development of Evidence based care in Heart disease Evaluated According to Recommended Therapies (SWEDEHEART) electronic data collection platform.

ELIGIBILITY:
Inclusion Criteria:

* Operated with minimally invasive mitral valve surgery between February 2016 and March 2019 at the Karolinska University Hospital in Stockholm, Sweden, with use of either surgical cut-down and arterial puncture under direct vision or percutaneously with planned percutaneous arteriotomy closed using a plug-based arteriotomy closure device.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patientes operated with minimally invasive mitral valve surgery between February 2016 and March 2019 at the Karolinska University Hospital in Stockholm, Sweden, with use of either surgical cut-down and arterial puncture under direct vision or percutaneously with planned percutaneous arteriotomy closed using a plug-based arteriotomy closure device.
Sampling Method: Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Major vascular groin-related complication according to the VARC-2 definition criteria | During the first 8 weeks after surgery

SECONDARY OUTCOMES:
Minor vascular groin-related complication according to the VARC-2 definition criteria | During the first 8 weeks after surgery
Access-site related groin seroma | During the first 8 weeks after surgery
Access-site related groin infection | During the first 8 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data not planned to be shared.

REFERENCES:
- [Derived] Kastengren M, Svenarud P, Kallner G, Settergren M, Franco-Cereceda A, Dalen M. Percutaneous Vascular Closure Device in Minimally Invasive Mitral Valve Surgery. Ann Thorac Surg. 2020 Jul;110(1):85-91. doi: 10.1016/j.athoracsur.2019.10.038. Epub 2019 Nov 30. PMID 31794742